CLINICAL TRIAL: NCT06004466
Title: The Development of Novel Noninvasive Internal Jugular Venous Oximetry
Brief Title: Noninvasive Internal Jugular Venous Oximetry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202203103DIND
Record Dates: First submitted 2023-08-17; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, we are developing a novel plethysmographic monitoring device which incorporates several key techniques: inclusion of structural information (ultrasound image), coupling with the estimation of local tissue optical parameters, consideration of the tissue scattering absorption coefficient of each subject, to finally calculate the noninvasive continuous internal jugular venous saturation.

DETAILED DESCRIPTION:
Central venous oxygen (ScvO2) is an important index for evaluating tissue perfusion in clinical care. To obtain the ScvO2 value, blood analysis must be obtained through a central venous catheter (CVC). Although CVC placement has a low incidence of complications, however, detrimental complications such as pneumothorax, hemothorax, infection and arrhythmia, are often fatal. In addition, continuous monitoring of ScvO2 often requires expensive equipment, so usually clinical caregivers can only take blood tests at specific care intervals, and may miss the opportunity to detect disease deterioration. In terms of anatomical structure and physiology, the values of internal jugular blood oxygen (SijvO2) and ScvO2 should be very close, and the evidence in the literature also points out that SijvO2 is not only highly similar to ScvO2, but also related to changes in cerebral blood oxygen. The internal jugular vein location is also an easier location for non-invasive continuous monitoring and thus it is interested to develop the novel technique for noninvasive continuous SijvO2 monitoring.

In this study, we are developing a novel plethysmographic monitoring device which incorporates several key techniques: inclusion of structural information (ultrasound image), coupling with the estimation of local tissue optical parameters, consideration of the tissue scattering absorption coefficient of each subject, to finally calculate the noninvasive continuous internal jugular venous saturation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing major cancer surgery that requires central venous catheter placement
* Cancer patients undergoing totally implantable venous access device placement

Exclusion Criteria:

* Susepct infectious symptoms and signs (eg. white blood cell count count >10000 ; fever >38.3℃)
* impaired liver functions (aspartate aminotransferase> 100 U/L); impaired renal function (estimated glomerular filtration rate <60 mL/min/1.73 m2)
* heart failure, with New York Heart Associatation class 2 or more

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cancer patients without organ dysfunction undergong planned central venous catheter placement for cancer surgery or totally implantable venous access device placement for future chemotherapy. During the central venous line placement, 3 ml blood sample from the internal jugular vein is obtained for internal validation of internal jugular venous saturation for our device.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Internal jugular venous saturation | 20 min
  To validate the estimation of noninvasive internal jugular venous saturation and the real value by obtaing the internal jugular venous blood during central venous catheter placement

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Yu Wu, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan